CLINICAL TRIAL: NCT03268785
Title: Intra-operative Rapid Identification of Lymph Node and Parathyroid by Fine Needle Puncture for Thyroid Carcinoma
Brief Title: Intra-operative Rapid Identification of Lymph Node and Parathyroid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Rui, Professor, Xijing Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20162049-X-1
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Thyroid Cancer; Parathyroid; Absent; Hypocalcemia; Hypoparathyroidism Postprocedural
Keywords: Parathyroid glands; Needle puncture; Diff-quik staining; PTH test assay; Thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Hypocalcemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Previous admitted patients who were given conventional thyroidectomy combined with central neck lymph node dissection, without intra-operative nodes identification were enrolled into control group.
- Experimental group (Experimental): Newly admitted patients,from august 2016 to august 2018, who were given thyroidectomy combined with central neck lymph node dissection, with intra-operative identification of suspicious lymph nodes or parathyroid glands were regarded as experimental group.Intraoperative identification method includes Diff-quik staining and PTH test assay. 200 participants were planed for enrollment.
  Interventions: Diagnostic Test: Intraoperative identification method

INTERVENTIONS:
Diagnostic Test: Intraoperative identification method — After needle pucture of suspicious nodes, Diff-quik staining was used to distinct lymph nodes and parathyroid glands. PTH test assay was used for parathyroid identification. Postoperative HE staining were applied as golden standard.
  Arms: Experimental group

SUMMARY:
During surgery, a fine needle puncture was proceeded when suspicious nodes was found by clinician. Repeat the punction for 2-3 times from different orientation and then, Diff-quik staining or PTH immunochromatographic assay were proceeded for lymph node or parathyroid glands identification. Post-operative pathology outcome was considered as golden standard.

DETAILED DESCRIPTION:
In the experiment group, when suspicious parathyroid glands or lymph nodes were observed, a 22 G needle was applied for in situ puncture at a 45 degree angle. The needle was initially thrust into the gland for 0.2 mm, and then we advanced the needle for another 0.2mm while gently withdrawing the plunger of the syringe and maintaining negative pressure. At this point, there has parathyroid tissue been adsorbed in the needle. Repeat this process in two different directions to guarantee the simple volume.

When cell smears finished, the smears were fixed in stationary liquid within 2-4 seconds for 5-20 seconds, and then Diff-Quik (DQ) staining technique was proceeded for rapid identification using Diff-Quik staining kit according to the instruction. After the following Diff-quick staining for 30 seconds, we can make out parathyroid cells and lymph nodes under high power microscope.

In addition,PTH immunochromatographic assay kit can also be used for parathyroid glands detection. Using indicator paper to dip to the punctured tissue, the existance of parathyroid glands could be ensured.

HE (Hematoxylin and Eosin) staining was used for pathological verification of suspicious nodes found during surgery. The suspicious nodes occurred in surgery were isolated and fixed with 4% paraformaldehyde for 12 h, embedded in parafﬁn and cut into 3-µm serial sections. Corresponding sections were stained with hematoxylin (BASO Diagnostics Inc. Zhuhai) for 10 min at room temperature. Then, sections were washed with running water. Subsequently, sections were washed with Scott promote blue liquid for 1 min, 1% hydrochloric acid alcohol differentiation liquid for 20 s, and Scott promote blue liquid for 1 min. Then, sections were stained with eosin (BASO Diagnostics Inc. Zhuhai) for 30 s. Sections were washed with running water and sealed for observation. Finally, sections were observed by Image-Pro Plus 5.0 software (Media Cybernetics, Inc., Bethesda, MD, USA).

ELIGIBILITY:
Inclusion Criteria:

- Thyroid cancer patients undergoing thyroid cancer surgery Preoperative examination were all ready for surgery Diagnosed with thyroid cancer by fine needle puncture before surgery

Exclusion Criteria:

- Patients enrolled into another clinical study Pregnant patients Patients diagnosed with another life-treating disease Patients with surgical contraindication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
hypocalcemia | 7 days after surgery
  Rate of hypocalcemia after surgery

SECONDARY OUTCOMES:
Accuracy,sensitivity and specificity | 10 day after operation
  Accuracy,sensitivity and specificity of intraoperative identification method
Life quality | 3 months after surgery
  The EORTC QLQ-C30 questionnaire was used to assess the life quality of participances. We calculate the score from 5 functional aspects according to the questionnnaire.
operation time | During the operation
  Record the identification time of this novel method and the whole operation time

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xijing hospital, Xi'an, Shaanxi
  - Xijing Hospital, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler JT, Sippel RS, Schaefer S, Chen H. Preserving function and quality of life after thyroid and parathyroid surgery. Lancet Oncol. 2008 Nov;9(11):1069-75. doi: 10.1016/S1470-2045(08)70276-6. PMID 19012855
- [Background] Carter Y, Chen H, Sippel RS. An intact parathyroid hormone-based protocol for the prevention and treatment of symptomatic hypocalcemia after thyroidectomy. J Surg Res. 2014 Jan;186(1):23-8. doi: 10.1016/j.jss.2013.09.026. Epub 2013 Oct 8. PMID 24144426
- See also: An intact parathyroid hormone-based protocol for the prevention and treatment of symptomatic hypocalcemia after thyroidectomy — https://www.ncbi.nlm.nih.gov/pubmed/?term=An+intact+parathyroid+hormone-based+protocol+for+the+prevention+and+treatment+of+symptomatic+hypocalcemia+after+thyroidectomy
- See also: Preserving function and quality of life after thyroid and parathyroid surgery. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Preserving+function+and+quality+of+life+after+thyroid+and+parathyroid+surgery